CLINICAL TRIAL: NCT05248464
Title: Association Between the Presence of Distress Related to the Feeling of Loss of Dignity and Quality of Life in Patients With Rheumatic Diseases
Brief Title: Distress Related to the Feeling of Loss of Dignity in Patients With Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Principal Investigator, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-4031-22/23-1
Record Dates: First submitted 2022-01-30; First posted 2022-02-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Rheumatic Diseases; Dignity; Quality of Life; Distress, Emotional
MeSH Terms: conditions — Rheumatic Diseases | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatic diseases patients: All the rheumatic diseases outpatients from the National Institute of Medical Sciences
  Interventions: Other: The Patient Dignity Inventory instrument (PDI); Other: WHOQOL-BREF (quality of life) instrument

INTERVENTIONS:
Other: The Patient Dignity Inventory instrument (PDI) — The PDI is an instrument made up of 25 items integrated into 5 factors that include: symptoms, existential anguish, dependency, peace of mind, and social support, prior to its application, adaptation, and validation will performer
Other: WHOQOL-BREF (quality of life) instrument — The WHOQOL-BREF is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment, it consists of 24 items.

SUMMARY:
Rheumatic diseases (RD) are an important group of different clinical entities and specific diseases that affect a significant proportion of the world population. In Mexico, the RD have a relevant representation in the adult population.

Dignity is a construct characterized by the representation of the self, of the self from others' point of view, and of the interaction of the individual with the environment and social context.

Living with a chronic illness can threaten experiences of dignity for the sick person and their families. Various studies have demonstrated the direct impact of the disease on dignity in terms of physical and psychological symptoms and loss of function. Some efforts have been made to operationalize the concept of perceived dignity in the context of chronic diseases

The perceived dignity of patients and the distress related to the feeling of loss of dignity (DRFLD) are outcomes that the patient can report and that the doctors can evaluate to be incorporated into the considerations of comprehensive care. Both outcomes are closely related, perceived dignity refers to a complex phenomenon, while distress related to the feeling of loss of dignity identifies those patients with a perceived dignity compromise of such magnitude that it generates anguish.

DETAILED DESCRIPTION:
The Patient Dignity Inventory (PDI) is an instrument originally written in English made up of 25 items integrated into 5 factors that include: symptoms, existential anguish, dependency, peace of mind and social support. Has a Likert-type response system with a 5-point scale, ranging from 1 ''not a problem'' to 5 ''very serious problem"; higher scores indicate greater dignity-related distress.

The PDI has been translated and validated into different languages, including validation in Spanish. The PDI instrument was validated in Mexico by Rodríguez-Mayoral et al., in 290 cancer patients. It had very good reliability with an alpha of 0.95 and a 4-factor structure that explained 64% of the variance (loss of meaning in life, loss of autonomy, dependency, and social support).

The primary objective of the study is the association between the presence of distress related to the feeling of loss of dignity and quality of life in patients with RD

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatic disease diagnosis according to their primary rheumatologist who agree to participate

Exclusion Criteria:

* Patients with a not confirmed rheumatic disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the rheumatic diseases from the National Institute of Medical Sciences and Nutrition
Sampling Method: Non-Probability Sample
Enrollment: 309 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence (percentage) of the presence of distress related to the feeling of loss of dignity in patients with RD | Baseline (At study inclusion)
  Determine the prevalence (percentage) of the presence of distress related to the feeling of loss of dignity in patients with RD, using PDI (distress related to the feeling of loss of dignity) instrument

SECONDARY OUTCOMES:
Determine the quality of life in patients with RD, using WHOQOL-BREF (quality of life) instrument | Baseline (At study inclusion)
  Determine the quality of life in patients with RD, using WHOQOL-BREF (quality of life) instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascual-Ramos V, Contreras-Yanez I, Cuevas-Montoya M, Guaracha-Basanez G, Garcia-Alanis M, Rodriguez-Mayoral O, Chochinov HM. The impact of underlying RMD diagnosis on dignity landscape in patients with systemic lupus erythematosus, rheumatoid arthritis, and systemic sclerosis. Medicine (Baltimore). 2025 Jul 18;104(29):e43303. doi: 10.1097/MD.0000000000043303. PMID 40696675